CLINICAL TRIAL: NCT02951962
Title: A Phase 1, Open Label, Two-cohort, Single-Sequence, Crossover Study to Investigate the Pharmacokinetic Drug Interaction and Safety of Telmisartan/Amlodipine and Rosuvastatin in Healthy Male Volunteers
Brief Title: A Study to Investigate Pharmacokinetic Drug Interaction and Safety of Telmisartan/Amlodipine and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP1604-101
Record Dates: First submitted 2016-08-21; First posted 2016-11-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — telmisartan amlodipine combination; Telmisartan; Amlodipine; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Twynsta 80/5mg (Experimental): Day 1 ~ Day 9 : Twynsta 80/5mg / Day 10 ~ Day 14 : Twynsta 80/5mg + Crestor 20mg
  Interventions: Drug: Twynsta 80/5mg; Drug: Crestor 20mg
- Crestor 20mg (Experimental): Day 1 ~ Day 5 : Crestor 20mg / Day 6 ~ Day 14 : Twynsta 80/5mg + Crestor 20mg
  Interventions: Drug: Twynsta 80/5mg; Drug: Crestor 20mg

INTERVENTIONS:
Drug: Twynsta 80/5mg — Hypertension
  Other Names: Telmisartan/Amlodipine 80/5mg
Drug: Crestor 20mg — Hyperlipidemia
  Other Names: Rosuvastatin 20mg

SUMMARY:
This is a phase 1, open label, two-cohort, single-sequence, crossover study

DETAILED DESCRIPTION:
This is a phase 1, open label, two-cohort, single-sequence, crossover study to investigate the pharmacokinetic drug interaction and safety of Telmisartan/Amlodipine and Rosuvastatin in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male with body mass index(BMI) between 18.5 and 28 kg/m2
* Who has not suffered from clinically significant disease
* Provision of signed written informed consent

Exclusion Criteria:

* History of and clinically significant disease
* A history of drug abuse or the presence of positive reactions to drugs that have abuse potential in urine screenings for drugs
* Administration of other investigational products within 3 months prior to the first dosing
* Volunteers considered not eligible for the clinical trial by the investigator due to reasons including laboratory test results, ECGs, or vital signs
* Sitting blood pressure meeting the following criteria at screening: 160 ≥ systolic blood pressure ≤100 (mmHg) and 95 ≥ diastolic blood pressure ≤ 60 (mmHg)

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Telmisartan, Amlodipine, Rosuvastatin AUCτ | 0 - 24 hr
Telmisartan, Amlodipine, Rosuvastatin Cmax | 0 - 24 hr

SECONDARY OUTCOMES:
Telmisartan, Amlodipine, Rosuvastatin Tmax | 0 - 24 hr
Telmisartan, Amlodipine, Rosuvastatin Cmin | 0 - 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No